CLINICAL TRIAL: NCT05097066
Title: Patterns and Outcomes of Neurosurgery in England Over a Five-year Period: a National Retrospective Cohort Study
Brief Title: Patterns and Outcomes of Neurosurgery in England Over a Five-year Period
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: The Royal College of Surgeons of England (Other)
Responsible Party: Principal Investigator, Ryan Mathew, Associate Professor and Consultant Neurosurgeon, University of Leeds
Other Study IDs: NNAP002
Record Dates: First submitted 2021-09-14; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Surgery; Surgery--Complications; Neurological Morbidity; Neurological Diseases or Conditions; Neurological Disorder; Neurological Complication; Neurological Procedural Complication; Outcome, Fatal; Comorbidities and Coexisting Conditions; Morality
MeSH Terms: conditions — Nervous System Diseases | interventions — Neurosurgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elective neurosurgery: Any elective neurosurgical procedure.
  Interventions: Procedure: Neurosurgical procedure
- Non-elective neurosurgery: Any non-elective neurosurgical procedure.
  Interventions: Procedure: Neurosurgical procedure

INTERVENTIONS:
Procedure: Neurosurgical procedure — Any neurosurgical procedure in the National Neurosurgical Audit Programme (NNAP) Coding Framework of neurosurgical procedures.

SUMMARY:
Neurosurgical practice has seen many important changes over several decades with advances in treatments and the types of patients treated. Neurosurgical procedures have evolved, and as outcomes have improved the number of patients being treated has increased.

There are no recent evaluations of national neurosurgical practice in the United Kingdom (UK), with the last prospective cohort studies being Safe Neurosurgery 1993 and Safe Neurosurgery 2000. More recent studies of neurosurgical services have been based on data from single institutions or surgeons and these may not give a representative picture of practice nationally.

Recent national quality improvement programmes for neurosurgery in England (such as the National Neurosurgical Audit Programme (NNAP) and Cranial Neurosurgery and Spinal Surgery Getting It Right First Time (GIRFT) Programmes) have focused on using national hospital administrative datasets. To be effective, quality improvement initiatives require robust outcome measures and quality (process) indicators. Currently, there is a lack of validated quality indicators for neurosurgery, with practice often being described using generic measures such as readmission and reoperation rates and length of stay. Many studies have been able to derive these common outcome measures, but it may also be possible to produce indicators specific to neurosurgery.

The aim of this observational study was firstly to describe the current pattern of neurosurgical admissions and procedures in England, and thereby given an overview of the epidemiology of neurosurgical patients. Secondly, it aims to investigate the range of outcome measures that might be produced from hospital administrative data and use these to assess the quality of care in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* All admissions to neurosurgical units in the National Health Service (NHS) in England.

Exclusion Criteria:

* Records with poor quality data (e.g. no data for clinical diagnoses).
* Patients under 18 years that were admitted to an adult neurosurgical unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All admissions to neurosurgical units in the National Health Service (NHS) in England. This covers any patients in England who required neurosurgical care, except those admitted to Private Providers of neurosurgical care.
Sampling Method: Non-Probability Sample
Enrollment: 371418 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | From date of admission to date of discharge from hospital; assessed up to 60 months.
  Length of the hospital admission to neurosurgery
Additional inpatient neurosurgical procedure rate | From date of admission to date of discharge from hospital; assessed up to 60 months.
  A further neurosurgical procedure in admissions where patients have had a primary (main) neurosurgical procedure.
Proportion of patients discharged home | Determined on date of discharge from hospital; assessed up to 60 months.
  Proportion of patients discharged to their normal address.
In-patient mortality rate | From date of the neurosurgical procedure through date of death from any cause (in-patient deaths only); assessed up to 60 months.
  In-patient mortality after a neurosurgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mathew, Study Chair — University of Leeds

IPD SHARING:
Plan to Share IPD: No